CLINICAL TRIAL: NCT06581016
Title: Performance Characteristics and Technical Outcomes of Single-use Versus Reusable Gastroscopes Evaluated in the Operating Room in Acute, Subacute and Elective Patients
Brief Title: Performance Characteristics and Technical Outcomes of Single-use vs. Reusable Gastroscopes Evaluated in the OR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zealand University Hospital (Other)
Collaborators: University Hospital, Umeå (Other)
Responsible Party: Principal Investigator, Camilla Kjelkvist-Born, Principal Investigator, Zealand University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SUSUES_COP
Record Dates: First submitted 2024-08-26; First posted 2024-08-30 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Upper Gastrointestinal Disorder
Keywords: Gastroscopy; Upper endoscopy; Gastroscope; Single-use; Reusable
MeSH Terms: conditions — Gastrointestinal Diseases

STUDY DESIGN:
Intervention Model Description: Non-inferiority, quality assurance study comparing a period where single-use gastroscopes are used with a period where reusable gastroscopes are used.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Single-use gastroscope (Experimental): In the first period all gastroscopies in the operating theater will be performed with single-use gastroscopes.
  Interventions: Device: Ambu aScope Gastro; Device: Ambu aScope Gastro Large
- Reusable gastroscope (Active Comparator): In the second period all gastroscopies in the operation theater will be performed with reusable gastroscopes.
  Interventions: Device: Diagnostic gastroscopes, Olympus; Device: Therapeutic gastroscopes, Olympus

INTERVENTIONS:
Device: Ambu aScope Gastro — CE-marked single-use gastroscopes from Ambu are used in the single-use group.
  Arms: Single-use gastroscope
Device: Ambu aScope Gastro Large — CE-marked single-use gastroscopes from Ambu are used in the single-use group.
  Arms: Single-use gastroscope
Device: Diagnostic gastroscopes, Olympus — Reusable gastroscopes from Olympus are used in the reusable group.
  Arms: Reusable gastroscope
Device: Therapeutic gastroscopes, Olympus — Reusable gastroscopes from Olympus are used in the reusable group.
  Arms: Reusable gastroscope

SUMMARY:
The goal of this clinical trial is to investigate whether single-use gastroscopes are as good as reusable gastroscopes when used in the operation theater in all patients where gastroscopy in the operation theater is indicated. The main question it aims to answer is:

- Is the technical success and performance characteristics the same for single-use and reusable gastroscopies?

Researchers will compare single-use gastroscopes with reusable gastroscopes to see if the technical success and performance characteristics are the same in the to groups.

Participants will in the first period have gastroscopy with a single-use gastroscope. In the second period participants will have gastroscopy with a reusable gastroscope.

ELIGIBILITY:
Inclusion Criteria:

* Acute, subacute or elective gastroscopies in the operating theater
* Age ≥ 18 years

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 700 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Technical success of single-use gastroscopes vs reusable gastroscopes | From admission to discharge, up to 3 months
  Technical success is defined as the ability to complete the procedure adequately based on the indication and guidelines.

SECONDARY OUTCOMES:
Complications | 24 hours and 72 hours follow-up after procedure
  Complications to gastroscopy
30th day mortality | 30 days
  Mortality after 30 days after procedure
Endoscopist's rating of gastroscope | Right after procedure
  The endoscopist's rating of the gastroscope
Duration of procedure | During the procedure
  The time from intubation of gastroscope until gastroscope removed from esophagus.
Time from procedure to discharge | From procedure to discharge, up to 3 months
  Time from procedure to discharge
Success of specific therapeutic procedures | During the procedure
  E.g. success in treating ulcers, banding or stenting
Need of new gastroscopy | During admission, up to 3 months
  Need of new gastroscopy during admission
Readmission | 30 days after procedure
  Does the patient need readmission after discharge
Sufficient ability to target the biopsy if taken | During procedure
  Successful biopsy which the pathologist can use to either diagnose the patient or to reject a diagnose.

CONTACTS AND LOCATIONS:
Overall Officials: Lasse Bremholm Hansen, PhD,ass.prof, Study Chair — Surgical department of Zealand University Hospital
Locations (1):
- Zealand University Hospital, Køge, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Turk DJ, Kozarek RA, Botoman VA, Patterson DJ, Ball TJ. Disposable endoscopic biopsy forceps: comparison with standard forceps of sample size and adequacy of specimen. J Clin Gastroenterol. 1991 Feb;13(1):76-8. PMID 2007750
- [Background] Forbes N, Elmunzer BJ, Allain T, Parkins MD, Sheth PM, Waddell BJ, Du K, Douchant K, Oladipo O, Saleem A, Cartwright S, Chau M, Howarth M, McKay J, Nashad T, Ruan Y, Bishay K, Gonzalez-Moreno E, Meng ZW, Bass S, Bechara R, Cole MJ, Jalink DW, Mohamed R, Turbide C, Belletrutti PJ, Kayal A, Kumar PR, Hilsden RJ, Buret AG, Hookey L, Heitman SJ. Effect of Disposable Elevator Cap Duodenoscopes on Persistent Microbial Contamination and Technical Performance of Endoscopic Retrograde Cholangiopancreatography: The ICECAP Randomized Clinical Trial. JAMA Intern Med. 2023 Mar 1;183(3):191-200. doi: 10.1001/jamainternmed.2022.6394. PMID 36689215
- [Background] Ross AS, Bruno MJ, Kozarek RA, Petersen BT, Pleskow DK, Sejpal DV, Slivka A, Moore D, Panduro K, Peetermans JA, Insull J, Rousseau MJ, Tirrell GP, Muthusamy VR. Novel single-use duodenoscope compared with 3 models of reusable duodenoscopes for ERCP: a randomized bench-model comparison. Gastrointest Endosc. 2020 Feb;91(2):396-403. doi: 10.1016/j.gie.2019.08.032. Epub 2019 Nov 1. PMID 31679738
- [Background] Bruno MJ, Beyna T, Carr-Locke D, Chahal P, Costamagna G, Devereaux B, Giovannini M, Goenka MK, Khor C, Lau J, May G, Muthusamy VR, Patel S, Petersen BT, Pleskow DK, Raijman I, Reddy DN, Repici A, Ross AS, Sejpal DV, Sherman S, Siddiqui UD, Ziady C, Peetermans JA, Rousseau MJ, Slivka A; EXALT Single-use Duodenoscope Study Group. Global prospective case series of ERCPs using a single-use duodenoscope. Endoscopy. 2023 Dec;55(12):1103-1114. doi: 10.1055/a-2131-7180. Epub 2023 Jul 18. PMID 37463599
- [Background] Ramai D, Smit E, Kani HT, Papaefthymiou A, Warner L, Chandan S, Dhindsa B, Facciorusso A, Gkolfakis P, Ofosu A, Barakat M, Adler DG. Cannulation rates and technical performance evaluation of commericially available single-use duodenoscopes for endoscopic retrograde cholangiopancreatography: A systematic review and meta-analysis. Dig Liver Dis. 2024 Jan;56(1):123-129. doi: 10.1016/j.dld.2023.02.022. Epub 2023 Mar 30. PMID 37003844
- [Background] Luo X, Ji M, Zhang S, Chen X, Zong Y, Zhang X, Hu H, Hao X, Shao L, Sun C, Shi H, Wang J, Wang B, Li P. Disposable versus reusable gastroscopes: a prospective randomized noninferiority trial. Gastrointest Endosc. 2022 Aug;96(2):250-261. doi: 10.1016/j.gie.2022.03.024. Epub 2022 Apr 4. PMID 35381230
- [Background] Li DF, Shi RY, Tian YH, Xu ZL, Zhou YS, Sun XJ, Cai JW, Fang YY, Peng H, Wang JM, Dong T, Cai YD, Yao J, Wang LS. The feasibility and safety of disposable endoscope vs. conventional endoscope for upper gastrointestinal tract examination: a multicenter, randomized, parallel, non-inferiority trial. Z Gastroenterol. 2022 Sep;60(9):1314-1319. doi: 10.1055/a-1555-0568. Epub 2021 Nov 12. PMID 34768288
- [Background] van der Ploeg K, de Jonge PJF, Lammers WJ, Koch AD, Vos MC, Paulsen V, Aabakken L, Bruno M. Performance of a single-use gastroscope for esophagogastroduodenoscopy: Prospective evaluation. Endosc Int Open. 2024 Mar 18;12(3):E428-E434. doi: 10.1055/a-2271-2303. eCollection 2024 Mar. PMID 38504741
- [Background] Ebigbo A, Tadic V, Schlottmann J, Braun G, Prinz F, Wanzl J, Ayoub M, Kraus L, Scheppach M, Nagl S, Schnoy E, Weber T, Probst A, Messmann H, Rommele C. Evaluation of a single-use gastroscope in patients presenting with suspected upper gastrointestinal hemorrhage: a pilot feasibility study (One-Scope I). Endoscopy. 2023 Oct;55(10):940-944. doi: 10.1055/a-2089-5969. Epub 2023 May 9. PMID 37160261
- [Background] Han ZL, Lin BT, Wang ZJ, Chen X, Xi YY, Wang JF, Qiao WG, Huang Y, Lin ZZ, Huang SH, Chua TY, Liu SD, Luo XB. Evaluation of a novel disposable esophagogastroduodenoscopy system in emergency, bedside, and intraoperative settings: Pilot study (with videos). Dig Endosc. 2023 Nov;35(7):857-865. doi: 10.1111/den.14548. Epub 2023 Apr 5. PMID 36905288
- [Background] Barakat MT, Banerjee S. Novel Algorithms for Reprocessing, Drying and Storing Endoscopes. Gastrointest Endosc Clin N Am. 2020 Oct;30(4):677-691. doi: 10.1016/j.giec.2020.06.003. Epub 2020 Jul 30. PMID 32891225
- [Background] Deb A, Perisetti A, Goyal H, Aloysius MM, Sachdeva S, Dahiya D, Sharma N, Thosani N. Gastrointestinal Endoscopy-Associated Infections: Update on an Emerging Issue. Dig Dis Sci. 2022 May;67(5):1718-1732. doi: 10.1007/s10620-022-07441-8. Epub 2022 Mar 9. PMID 35262904
- [Background] Larsen S, Kalloo A, Hutfless S. The hidden cost of colonoscopy including cost of reprocessing and infection rate: the implications for disposable colonoscopes. Gut. 2020 Feb;69(2):197-200. doi: 10.1136/gutjnl-2019-319108. Epub 2019 Aug 14. No abstract available. PMID 31413166
- [Background] Bang JY, Sutton B, Hawes R, Varadarajulu S. Concept of disposable duodenoscope: at what cost? Gut. 2019 Nov;68(11):1915-1917. doi: 10.1136/gutjnl-2019-318227. Epub 2019 Feb 12. No abstract available. PMID 30772837
- [Background] Cennamo V, Botter A, Landi S, Graziosi F, Bassi M, Dabizzi E, Ghersi S, Cerone G, Bonfiglioli R. Can single-use versus standard duodenoscope improve ergonomics in ERCP? A comparative, simulation-based pilot study. Endosc Int Open. 2024 Mar 18;12(3):E419-E427. doi: 10.1055/a-2231-7393. eCollection 2024 Mar. PMID 38504744
- [Background] Le NNT, Hernandez LV, Vakil N, Guda N, Patnode C, Jolliet O. Environmental and health outcomes of single-use versus reusable duodenoscopes. Gastrointest Endosc. 2022 Dec;96(6):1002-1008. doi: 10.1016/j.gie.2022.06.014. Epub 2022 Jun 17. PMID 35718068
- [Background] Namburar S, von Renteln D, Damianos J, Bradish L, Barrett J, Aguilera-Fish A, Cushman-Roisin B, Pohl H. Estimating the environmental impact of disposable endoscopic equipment and endoscopes. Gut. 2022 Jul;71(7):1326-1331. doi: 10.1136/gutjnl-2021-324729. Epub 2021 Dec 1. PMID 34853058
- [Background] Rodriguez de Santiago E, Dinis-Ribeiro M, Pohl H, Agrawal D, Arvanitakis M, Baddeley R, Bak E, Bhandari P, Bretthauer M, Burga P, Donnelly L, Eickhoff A, Hayee B, Kaminski MF, Karlovic K, Lorenzo-Zuniga V, Pellise M, Pioche M, Siau K, Siersema PD, Stableforth W, Tham TC, Triantafyllou K, Tringali A, Veitch A, Voiosu AM, Webster GJ, Vienne A, Beilenhoff U, Bisschops R, Hassan C, Gralnek IM, Messmann H. Reducing the environmental footprint of gastrointestinal endoscopy: European Society of Gastrointestinal Endoscopy (ESGE) and European Society of Gastroenterology and Endoscopy Nurses and Associates (ESGENA) Position Statement. Endoscopy. 2022 Aug;54(8):797-826. doi: 10.1055/a-1859-3726. Epub 2022 Jul 8. PMID 35803275
- [Background] Mackiewicz-Pracka A, Nehring P, Przybylkowski A. Emergency Endoscopic Interventions in Acute Upper Gastrointestinal Bleeding: A Cohort Study. Diagnostics (Basel). 2023 Dec 1;13(23):3584. doi: 10.3390/diagnostics13233584. PMID 38066825
- See also: US Food and Drug Administration. News & Events; FDA Newsroom; Press Announcements. FDA Continues Efforts to Support Innovation in Medical Device Sterilization (August 3, 2022). Accessed: 21 July 2023. — http://public4.pagefreezer.com/content/FDA/07-09-2023T11:58/https://www.fda.gov/news-events/press-announcements/fda-continues-efforts-support-innovation-medical-device-sterilization
- See also: Sealed Envelope Ltd. 2012. Power calculator for binary outcome non-inferiority trial. [Accessed Fri Jul 05 2024]. — http://www.sealedenvelope.com/power/binary-noninferior/